CLINICAL TRIAL: NCT03985709
Title: Deciphering the Role of the Microbiota in Osteoarthritis for Improving Therapy
Brief Title: Probiotic for Osteoarthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Responsible Party: Principal Investigator, Jorge Hugo Villafañe, PhD, Researcher, Fondazione Don Carlo Gnocchi Onlus
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Probiotic in OA
Record Dates: First submitted 2019-06-10; First posted 2019-06-14 (Actual); Last update posted 2019-06-14 (Actual); Status verified 2019-06

CONDITIONS: Osteoarthritis of Multiple Joints
Keywords: Osteoarthritis; Microbiota; Probiotic
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Probiotcal group (Experimental): Probiotic (Lactobacillus casei) once daily taken by 3 months
  Interventions: Other: Probiotic product

INTERVENTIONS:
Other: Probiotic product — Probiotic (Lactobacillus casei) once daily taken by 3 months.

SUMMARY:
The gut microbiome appears to be a significant contributor to musculoskeletal health and disease. Microbiome composition and its functional implications have been associated with prevention of bone loss and/or reducing fracture risk. Genetic background, gender, dietary intake, and social factors are also important factors which contribute to the musculoskeletal health, as well as to the normal balance of intestinal microbiota. The link between gut microbiota and joint inflammation in murine models of arthritis has been established, and it is now receiving increasing attention in human studies. Recent papers have demonstrated substantial alterations in the gut microbiota in patients with rheumatoid arthritis (RA) and osteoarthritis (OA). These alterations resemble those established in systemic inflammatory conditions (inflammatory bowel disease, spondyloarthritides, psoriasis), which include decreased microbial diversity and lower abundances of bacteria belonging to the Firmicutes phylum that are known to have immunoregulatory properties.These new findings open important future horizons both for understanding disease pathophysiology and for developing novel biomarkers and treatment strategies. Further investigation into the mechanisms linking changes in the microbiome to alterations in bones and joints is necessary. Next Generation Sequencing, metatranscriptomic analysis, and metabolomic approaches may provide yet-greater insight and help further understand these mechanisms. To investigate gut microbiota change will be associated with the sintoms of knee and / or hip OA in italian patients.

ELIGIBILITY:
Inclusion Criteria:

* All subjects will have hip or knee OA according on radiographic findings (Kellgren-Lawrence scale ≥3). A physiatrist (physician) will establish the diagnosis of pain-OA.

Exclusion Criteria:

* Psychiatric or neurological disorders, celiac disease, lactose intolerance, or allergies or other ongoing illnesses (i.e., irritable bowel syndrome, diabetes, ulcerative colitis, etc.) or recent antibiotic treatment (i.e., <3 months before the beginning of the study).
* Participants require treatment with aspirin > 325 mg /day.
* Participants who smoked more than 10 cigarettes per day were excluded.
* Participants will be excluded also if they score greater than 6 points on the Beck Depression Inventory (BDI) or more than 30 points in the State Trait Anxiety Inventory (STAI), dementia and not Italian speaking due to the high level of language skills required for questionnaires and quantitative sensory testing.
* Post-traumatic OA (e.g., fractures), congenital hip deformities, surgical interventions to the hip or knee, Legg-Calvé-Perthes disease, or degenerative or non-degenerative neurological conditions in which pain perception is altered will be excluded

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-02-01 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
Change from Pain Intensity at 3 months. | Baseline, immediately post-intervention (3 months).
  Visual Analogue Scale, 0: no pain, 100: maximum pain
Change from range of Pressure Pain Thresholds at 3 months | Baseline, immediately post-intervention (3 months).
  Algometry, will be assessed bilaterally [in the center of the anterior aspect of patella (knee) and the trochanter site (hip). The range of values of the pressure algometer was 0 to 10 kg.

SECONDARY OUTCOMES:
Change from concentrations of Inflammatory cytokines at 3 months. | Baseline, immediately post-intervention (3 months).
  Fasting serum concentrations of interleukin (IL)-6, tumor necrosis factor (TNF)-α, soluble IL-6 receptor (IL-6sR), soluble IL-1 receptor (IL-1sR), and C-reactive protein (CRP) were measured by enzyme-linked immunosorbent assays. All samples were measured in duplicate, and the average of the two values was used for data analyses.
Change from Microbiota at 3 months. | Baseline, immediately post-intervention (3 months).
  Microbiota composition will be identified through fecal samples for total genomic DNA extraction. The bacteria belonging to Clostridium sensu stricto, Enterobacteriaceae, Escherichia coli, Bifidobacterium, Lactobacillus and yeast were dosed using quantitative PCR approach targeted on 16S rRNA gene.

CONTACTS AND LOCATIONS:
Overall Officials: Jorge H Villafañe, PhD, Principal Investigator — Fondazione Don Carlo Gnocchi Onlus
Locations (1):
- Jorge Hugo Villafañe, Milan, Italy

IPD SHARING:
Plan to Share IPD: No